CLINICAL TRIAL: NCT06823791
Title: Efficacy and Safety of Furazolidone Containing Quadruple Therapy for First-line Helicobacter Pylori Eradication
Brief Title: Furazolidone Quadruple Regimen Eradicate H. Pylori Infection
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Liaocheng People's Hospital (Other)
Responsible Party: Principal Investigator, liulifeng, deputy chief doctor, Liaocheng People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1234567
Record Dates: First submitted 2023-09-04; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Helicobacter Pylori Infection; Eradication
Keywords: H. pylori eradication; furazolidone quadruple regimen; clarithromycin quadruple regimen
MeSH Terms: interventions — Furazolidone; Esomeprazole; Amoxicillin; Clarithromycin

STUDY DESIGN:
Intervention Model Description: A total of 500 patients with primary H pylori infection were collected from Liaocheng People's Hospital. Patients were randomly divided into FZD group and CLA group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- furazolidone regimen (Experimental): Patients who were enrolled in the experimental group use the furazolidone regimen esomeprazole magnesium 20 mg bid +colloidal bismuth pectin 200mg bid+ amoxicillin 1000 mg bid+ furazolidone 100 mg bid
  Interventions: Drug: Furazolidone
- Clarithromycin regimen (Active Comparator): Patients who were enrolled in the control group use the clarithromycin regimen esomeprazole magnesium 20 mg bid+colloidal bismuth pectin 200mg bid+ amoxicillin 1000 mg bid+ clarithromycin 500 mg bid
  Interventions: Drug: Clarithromycin

INTERVENTIONS:
Drug: Furazolidone — esomeprazole magnesium 20 mg bid +colloidal bismuth pectin 200mg bid + amoxicillin 1000 mg bid + furazolidone 100 mg bid, for 14 days. After stopping the medication for 30 days, check the H. pylori again. If H. pylori is negative, check again after 6 months and 12 months, the experiment stop. If H. pylori is positive, check again after 6 months. If H. pylori is still positive, high-dose dual therapy will be used to resist H. pylori again. After stopping the second medication for 30 days, check the H. pylori again. If H. pylori is negative, check again after 6 months, and the experiment stops. If H. pylori is still positive, check again after 6 months, and the experiment stops.
  Other Names: esomeprazole magnesium; colloidal bismuth pectin; amoxicillin
  Arms: furazolidone regimen
Drug: Clarithromycin — esomeprazole magnesium 20 mg bid +colloidal bismuth pectin 200mg bid + amoxicillin 1000 mg bid + clarithromycin 500 mg bid, for 14 days. After stopping the medication for 30 days, check the H. pylori again. If H. pylori is negative, check again after 6 months and 12 months, the experiment stop. If H. pylori is positive, check again after 6 months. If H. pylori is still positive, high-dose dual therapy will be used to resist H. pylori again. After stopping the second medication for 30 days, check the H. pylori again. If H. pylori is negative, check again after 6 months, and the experiment stops. If H. pylori is still positive, check again after 6 months, and the experiment stops.
  Other Names: esomeprazole magnesium; colloidal bismuth pectin; amoxicillin
  Arms: Clarithromycin regimen

SUMMARY:
Research protocol:

Experimental group:

First line solution (furazolidone regimen): esomeprazole magnesium 20 mg +colloidal bismuth pectin 200mg+ amoxicillin 1000 mg + furazolidone 100 mg, twice daily, for 14 days.

Patients who is still positive for H. pylori infection after the first line solution select the second line solution (high-dose dual regimen): esomeprazole magnesium 20 mg and amoxicillin 750 mg, 4 times daily, for 14 days.

Control group:

First line solution (clarithromycin regimen): esomeprazole magnesium 20 mg +colloidal bismuth pectin 200mg+ amoxicillin 1000 mg + clarithromycin 500 mg, twice a day, for 14 days.

Patients who is still positive for H. pylori infection after the first line solution select the second line solution (high-dose dual regimen): esomeprazole magnesium 20 mg and amoxicillin 750 mg, 4 times daily, for 14 days.

Main study endpoint:

The difference in the eradication rate of H. pylori infection between the furazolidone quadruple regimen and the clarithromycin quadruple regimen.

Secondary study endpoint:

1. Safety and compliance of the furazolidone quadruple regimen.
2. Comparison of high-dose dual therapy with furazolidone quadruple therapy and clarithromycin quadruple therapy on H. pylori eradication rate.
3. 1-year recurrence and recurrence rate of H. pylori infection.

DETAILED DESCRIPTION:
Patients A total of 500 patients with primary H pylori infection were collected from Liaocheng People's Hospital from August 2022 to July 2024. These patients were from outpatient clinics, followed up by using telephone to monitor drugs, adverse reactions, symptom improvement before and after medication. Written informed consent was obtained from all participated patients in this study. This study was approved by the local research ethics committee at the Liaocheng Hospital according to the principle of the Helsinki Declaration II (No. 2023110). Patients were randomly divided into FZD group and CLA group. Inclusion criteria include: 1. Hp test positive. 2. age range from 18 to 70 years. 3. without previously Hp eradication treatment prior to enrollment. Exclusion criteria were as follows: 1. severe concomitant diseases such as cardiac dysfunction, liver, kidney et al. 2. planning to be or being pregnant, or lactating. 3. history of allergy to any medicines used in this study. 4. lost in follow-up.

Drugs Drugs used in this study were as follows: FZD was from Shanghai Yurui Biotechnology Pharmaceutical Co., Ltd. Esomeprazole was from AstraZeneca Pharmaceutical Co. Ltd, England; AMX was from Shandong LuKang Pharmaceutical Co., Ltd; Bismuth potassium citrate was from Shanghai Modern Hassen Pharmaceutical Co., Ltd. CLA was from Guangdong DongYangGuang Pharmaceutical Co., Ltd. All drugs were routinely prescribed in hospital pharmacy.

Determination of Hp infection The status of Hp infection was determined by methods as follows: 1. 13C/14C urea breath test (UBT) 2. rapid urease test (RUT) 3. HE staining of gastric mucosal histopathological sections 4. gastric mucosal Hp culture 5. fecal Hp antigen test. Post-treatment Hp status was assessed 4 weeks after ﬁnishing the treatment. Hp was considered eradicated if post-treatment Hp was negative. If the result was positive, it was retested again after half a year. If the retested result was still positive, Hp eradication failed.

Hp eradication regimens and duration Patients were randomly allocated into FZD and CLA groups. The FZD group includes FZD (100mg, bid), esomeprazole (20mg, bid), bismuth potassium citrate (220mg, bid), and AMX (1000mg, bid) for 14 days. In the CLA group, FZD was replaced by CLA (500mg, bid), and the other drugs were the same. Esomeprazole and bismuth were taken 30 minutes before meal, AMX, CLA, and FZD were taken 30 minutes after meal.

Evaluation of adverse effects and symptom improvement after treatment Drugs, adverse effects, improvement of clinical symptoms were recorded by outpatient questionnaire. Adverse drug reactions include abdominal pain, bloating, diarrhea, constipation, nausea, changes in taste (bad oral taste), rash, insomnia, arthralgia, headache, dizziness, fatigue, peripheral nerve damage. The adverse events were classiﬁed as yes or no. The symptoms before and after treatment was evaluated by the Likert rating scale. Symptoms are classified as none (1 point), mild (2 points, almost no symptoms), moderate (3 points, tolerable, not affect daily activities), severe (4 points, affect daily activities), and serious (5 points, need to be hospitalized or intervened to prevent permanent injury or even death). Frequency includes: none (1 point), less than 2 times a week (2 points), more than 3 times a week and not daily (3 points), daily but intermittent (4 points), almost constant daily (5 points). Total score = frequency×symptom.

Cost-effectiveness analysis Cost (C) is the total cost of each regimen of drugs. Effectiveness (E) represents therapeutic effect of a regimen. In this study, cost-effectiveness ratio (C/E) and incremental cost-effectiveness ratio were used to evaluate the cost-effectiveness analysis. Incremental cost-effectiveness ratio (DC/DE) referred to the ratio of cost difference to effectiveness between FZD group and CLA group; which means the cost of each unit effect increased by former scheme.

ELIGIBILITY:
Inclusion Criteria:

1. H Pylori infection: 13C/14C urea breath test positive or rapid urease test positive or gastric mucosal tissue pathological section HE staining positive or gastric mucosal tissue H. Pylori culture positive or fecal Positive detection of H pylori antigen
2. No previous History of eradication treatment for H pylori;
3. Age 18-70 years old;

Exclusion Criteria:

1. Pregnant or lactating women;
2. There are also other serious diseases that affect the evaluation of this study, such as severe coronary heart disease, liver disease, kidney disease, chronic obstructive pulmonary disease, malignant tumors, and psychological disorders;
3. Individuals with a history of significant or complex gastrointestinal surgery;
4. Individuals who are allergic to the drugs used in this study;
5. Unable to cooperate with this experimenter.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 493 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Hp eradication rate | 6 months
  The status of Hp infection was determined by methods as follows: 1. 13C/14C urea breath test (UBT) 2. rapid urease test (RUT) 3. HE staining of gastric mucosal histopathological sections 4. gastric mucosal Hp culture 5. fecal Hp antigen test. Post-treatment Hp status was assessed 4 weeks after ﬁnishing the treatment. Hp was considered eradicated if post-treatment Hp was negative. If the result was positive, it was retested again after half a year. If the retested result was still positive, Hp eradication failed.

SECONDARY OUTCOMES:
adverse reactions | 1 month
  adverse effect was recorded by outpatient questionnaire. Adverse reactions include abdominal pain, abdominal distension, diarrhea, constipation, nausea, changes in taste (bad oral breath), rash, insomnia, arthralgia, headache, dizziness, fatigue, peripheral nerve damage.

CONTACTS AND LOCATIONS:
Overall Officials: Lifeng Liu, Principal Investigator — Liaocheng Peoples hospital
Locations (1):
- Liaocheng Peoples hospital, Liaocheng, Shandong, China

IPD SHARING:
Plan to Share IPD: No